CLINICAL TRIAL: NCT04358562
Title: A Randomized Phase II Trial of Gefitinib With Anlotinib in Advanced Non-squamous NSCLC Patients With Uncleared Plasma ctDNA EGFRm After First-line Treatment With Gefitinib
Brief Title: Gefitinib With Anlotinib in Advanced Non-squamous NSCLC Patients With Uncleared Plasma ctDNA EGFRm After First-line Treatment With Gefitinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20171BCD40022
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer; EGFR Gene Mutation
Keywords: Gefitinib; Anlotinib; EGFR Gene Mutation; Non-small Cell Lung Cancer; TKIs; Antivascular therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; anlotinib

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefitinib with Anlotinib (Experimental): If persistence of plasma ctDNA EGFRm after 8 weeks of gefitinib first-line treatment, Gefitinib 250mg oral daily and Anlotinib 10mg oral d1-14, every 3 weeks
  Interventions: Drug: Gefitinib; Drug: Anlotinib
- Gefitinib (Experimental): If clearance of plasma ctDNA EGFRm after 8 weeks of gefitinib first-line treatment, Gefitinib 250mg oral daily
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — If persistence of plasma ctDNA EGFRm after 8 weeks of gefitinib first-line treatment
  Other Names: Iressa
Drug: Anlotinib — If clearance of plasma ctDNA EGFRm after 8 weeks of gefitinib first-line treatment
  Other Names: AL3818
  Arms: Gefitinib with Anlotinib

SUMMARY:
TKIs therapy is the first-line treatment of patients with EGFR mutation advanced NSCLC.However, some patients have poor prognosis of drug resistance in the early stage. The dynamic alterations of ctDNA-based EGFR mutation after TKIs treatment is a predictor of the efficacy of TKIs treatment, which can be used to identify this part of patients in the early stage.Drug resistance can be overcome when TKIs is combined with drugs in different mechanisms of action, such as chemotherapy and anti-angiogenesis therapy.Gefitinib is the first-generation oral EGFR TKIs. Anlotinib is a domestic oral small molecule inhibitor of multireceptor tyrosine kinase, which has extensive inhibitory effect on tumor angiogenesis and growth.Gefitinib combined with anlotinib is a new option in the treatment of patients with uncleared plasma EGFRm after gefitinib treatment.

DETAILED DESCRIPTION:
This is an open-label, prospective, randomized, controlled phase II clinical trial.To evaluate the efficacy and safety of gefitinib combined with anlotinib versus gefitinib alone in advanced non-squamous NSCLC patients whose EGFRm was not cleared in plasma ctDNA after 8 weeks of gefitinib first-line treatment, so as to provide clinical basis for a new and tolerable treatment that can prolong the survival time of patients with advanced NSCLC. Study therapy continued until disease progression, unacceptable adverse event, or withdrawal of consent. The efficacy and adverse reactions of the trial regimen will be evaluated according to RECIST criteria and NCI-CTC AE V3.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed that EGFR sensitive mutation (ex19del or L858R mutation) in tumor tissue was detected by non-squamous NSCLC, and EGFR mutation (ex19del or L858R mutation) in ctDNA before treatment;
* Staging is IVB stage (AJCC 8th Edition) ;
* According to the comprehensive judgment of many disciplines, it is impossible to be treated by operation;
* PS score 0-1;
* The patient has at least one measurable tumor injury (the tumor is considered unmeasurable at the site of previous radiotherapy);
* Systemic anti-tumor therapy such as chemotherapy, immunotherapy and targeted therapy were not performed before entering the group;
* There is no history of malignant tumor and no serious medical disease;
* FEV1 ≥ 1.2L/ seconds or ≥ 50% predicted value;
* Laboratory examination: White blood cell count ≥ 4 *10^9/L, neutrophil count ≥ 2.0 *10^9, platelet count ≥ 100 *10^9, hemoglobin ≥ 10 g / L, liver and kidney function and ECG were normal;
* The pregnancy test was negative within 3 days before entering the group, and agreed to use medically effective contraceptive measures during the trial;
* Life expectancy is more than 12 weeks;
* Sign informed consent form; cooperate with regular follow-up.

Exclusion Criteria:

* T4 (AJCC 8th Edition) patients with severe destruction and stenosis of large vessels confirmed by imaging;
* Clinical severe infection (> grade 2 NCI-CTC V3.0);
* Severe immunosuppressive disease;
* The patient's physical condition is life-threatening;
* A pregnant or breastfeeding patient. Female patients who are likely to become pregnant must be tested negative within 7 days of the start of treatment before continuing. Patients enrolled in the trial (both male and female) must use contraception during the trial period until two weeks after the trial is completed;
* PS score ≥ 2;
* At the same time, there are other serious diseases (congestive heart failure, transmural myocardial infarction, COPD or other respiratory diseases that affect treatment, etc.), considering that the study may aggravate or fail to control the disease;
* Those who have suffered or are currently suffering from tumors whose primary site or histology are different from those evaluated in this study. Excluding cervical carcinoma in situ, cured basal cell carcinoma, bladder surface tumor [Ta,Tis&T1], or any cured tumor that has been in the study for more than 3 years;
* The patient refused to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival, PFS | Every 6 weeks up to 2 years
  The period from the start of treatment to the progression or death of a patient

SECONDARY OUTCOMES:
overall survival, OS | Every 6 weeks up to 2 years, and then every 3 months up to 5 years
  time from the beginning of study to death due to any cause or last follow-up
Objective Response Rate, ORR | 6 weeks after treatment
  ORR, proportion of patients with a best overall response of complete response or partial response (CR+PR)
adverse events | Every 6 weeks up to 2 years
  Number of patients with adverse events (AEs) as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Liu Anwen, Phd, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ke EE, Zhou Q, Wu YL. Emerging paradigms in targeted treatments for Asian patients with NSCLC. Expert Opin Pharmacother. 2015 Jun;16(8):1167-76. doi: 10.1517/14656566.2015.1040391. Epub 2015 Apr 23. PMID 25907450
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Domvri K, Zarogoulidis P, Darwiche K, Browning RF, Li Q, Turner JF, Kioumis I, Spyratos D, Porpodis K, Papaiwannou A, Tsiouda T, Freitag L, Zarogoulidis K. Molecular Targeted Drugs and Biomarkers in NSCLC, the Evolving Role of Individualized Therapy. J Cancer. 2013 Nov 23;4(9):736-54. doi: 10.7150/jca.7734. PMID 24312144
- [Result] Rosell R, Moran T, Queralt C, Porta R, Cardenal F, Camps C, Majem M, Lopez-Vivanco G, Isla D, Provencio M, Insa A, Massuti B, Gonzalez-Larriba JL, Paz-Ares L, Bover I, Garcia-Campelo R, Moreno MA, Catot S, Rolfo C, Reguart N, Palmero R, Sanchez JM, Bastus R, Mayo C, Bertran-Alamillo J, Molina MA, Sanchez JJ, Taron M; Spanish Lung Cancer Group. Screening for epidermal growth factor receptor mutations in lung cancer. N Engl J Med. 2009 Sep 3;361(10):958-67. doi: 10.1056/NEJMoa0904554. Epub 2009 Aug 19. PMID 19692684
- [Result] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Result] Schuler M, Tan EH, O'Byrne K, Zhang L, Boyer M, Mok T, Hirsh V, Yang JC, Lee KH, Lu S, Shi Y, Kim SW, Laskin J, Kim DW, Arvis CD, Kolbeck K, Massey D, Marten A, Paz-Ares L, Park K. First-line afatinib vs gefitinib for patients with EGFR mutation-positive NSCLC (LUX-Lung 7): impact of afatinib dose adjustment and analysis of mode of initial progression for patients who continued treatment beyond progression. J Cancer Res Clin Oncol. 2019 Jun;145(6):1569-1579. doi: 10.1007/s00432-019-02862-x. Epub 2019 Feb 19. PMID 30783814
- [Result] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Result] Pao W, Chmielecki J. Rational, biologically based treatment of EGFR-mutant non-small-cell lung cancer. Nat Rev Cancer. 2010 Nov;10(11):760-74. doi: 10.1038/nrc2947. Epub 2010 Oct 22. PMID 20966921
- [Result] Wu YL, Saijo N, Thongprasert S, Yang JC, Han B, Margono B, Chewaskulyong B, Sunpaweravong P, Ohe Y, Ichinose Y, Yang JJ, Mok TS, Young H, Haddad V, Rukazenkov Y, Fukuoka M. Efficacy according to blind independent central review: Post-hoc analyses from the phase III, randomized, multicenter, IPASS study of first-line gefitinib versus carboplatin/paclitaxel in Asian patients with EGFR mutation-positive advanced NSCLC. Lung Cancer. 2017 Feb;104:119-125. doi: 10.1016/j.lungcan.2016.11.022. Epub 2016 Nov 30. PMID 28212993
- [Result] Mitsudomi T, Morita S, Yatabe Y, Negoro S, Okamoto I, Tsurutani J, Seto T, Satouchi M, Tada H, Hirashima T, Asami K, Katakami N, Takada M, Yoshioka H, Shibata K, Kudoh S, Shimizu E, Saito H, Toyooka S, Nakagawa K, Fukuoka M; West Japan Oncology Group. Gefitinib versus cisplatin plus docetaxel in patients with non-small-cell lung cancer harbouring mutations of the epidermal growth factor receptor (WJTOG3405): an open label, randomised phase 3 trial. Lancet Oncol. 2010 Feb;11(2):121-8. doi: 10.1016/S1470-2045(09)70364-X. Epub 2009 Dec 18. PMID 20022809
- [Result] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Result] Gray JE, Okamoto I, Sriuranpong V, Vansteenkiste J, Imamura F, Lee JS, Pang YK, Cobo M, Kasahara K, Cheng Y, Nogami N, Cho EK, Su WC, Zhang G, Huang X, Li-Sucholeiki X, Lentrichia B, Dearden S, Jenkins S, Saggese M, Rukazenkov Y, Ramalingam SS. Tissue and Plasma EGFR Mutation Analysis in the FLAURA Trial: Osimertinib versus Comparator EGFR Tyrosine Kinase Inhibitor as First-Line Treatment in Patients with EGFR-Mutated Advanced Non-Small Cell Lung Cancer. Clin Cancer Res. 2019 Nov 15;25(22):6644-6652. doi: 10.1158/1078-0432.CCR-19-1126. Epub 2019 Aug 22. PMID 31439584
- [Result] Mok T, Wu YL, Lee JS, Yu CJ, Sriuranpong V, Sandoval-Tan J, Ladrera G, Thongprasert S, Srimuninnimit V, Liao M, Zhu Y, Zhou C, Fuerte F, Margono B, Wen W, Tsai J, Truman M, Klughammer B, Shames DS, Wu L. Detection and Dynamic Changes of EGFR Mutations from Circulating Tumor DNA as a Predictor of Survival Outcomes in NSCLC Patients Treated with First-line Intercalated Erlotinib and Chemotherapy. Clin Cancer Res. 2015 Jul 15;21(14):3196-203. doi: 10.1158/1078-0432.CCR-14-2594. Epub 2015 Mar 31. PMID 25829397
- [Result] Wang Z, Cheng Y, An T, Gao H, Wang K, Zhou Q, Hu Y, Song Y, Ding C, Peng F, Liang L, Hu Y, Huang C, Zhou C, Shi Y, Zhang L, Ye X, Zhang M, Chuai S, Zhu G, Hu J, Wu YL, Wang J. Detection of EGFR mutations in plasma circulating tumour DNA as a selection criterion for first-line gefitinib treatment in patients with advanced lung adenocarcinoma (BENEFIT): a phase 2, single-arm, multicentre clinical trial. Lancet Respir Med. 2018 Sep;6(9):681-690. doi: 10.1016/S2213-2600(18)30264-9. Epub 2018 Jul 17. PMID 30017884
- [Result] Lee CK, Brown C, Gralla RJ, Hirsh V, Thongprasert S, Tsai CM, Tan EH, Ho JC, Chu da T, Zaatar A, Osorio Sanchez JA, Vu VV, Au JS, Inoue A, Lee SM, Gebski V, Yang JC. Impact of EGFR inhibitor in non-small cell lung cancer on progression-free and overall survival: a meta-analysis. J Natl Cancer Inst. 2013 May 1;105(9):595-605. doi: 10.1093/jnci/djt072. Epub 2013 Apr 17. PMID 23594426
- [Result] Noronha V, Patil VM, Joshi A, Menon N, Chougule A, Mahajan A, Janu A, Purandare N, Kumar R, More S, Goud S, Kadam N, Daware N, Bhattacharjee A, Shah S, Yadav A, Trivedi V, Behel V, Dutt A, Banavali SD, Prabhash K. Gefitinib Versus Gefitinib Plus Pemetrexed and Carboplatin Chemotherapy in EGFR-Mutated Lung Cancer. J Clin Oncol. 2020 Jan 10;38(2):124-136. doi: 10.1200/JCO.19.01154. Epub 2019 Aug 14. PMID 31411950
- [Result] Ciardiello F, Bianco R, Damiano V, Fontanini G, Caputo R, Pomatico G, De Placido S, Bianco AR, Mendelsohn J, Tortora G. Antiangiogenic and antitumor activity of anti-epidermal growth factor receptor C225 monoclonal antibody in combination with vascular endothelial growth factor antisense oligonucleotide in human GEO colon cancer cells. Clin Cancer Res. 2000 Sep;6(9):3739-47. PMID 10999768
- [Result] Bozec A, Sudaka A, Fischel JL, Brunstein MC, Etienne-Grimaldi MC, Milano G. Combined effects of bevacizumab with erlotinib and irradiation: a preclinical study on a head and neck cancer orthotopic model. Br J Cancer. 2008 Jul 8;99(1):93-9. doi: 10.1038/sj.bjc.6604429. Epub 2008 Jun 24. PMID 18577994